CLINICAL TRIAL: NCT04884932
Title: Percutaneous High Frequency Alternating Current Stimulation: Effects on Somatosensory and Motor Threshold in Healthy Volunteers With 30 kHz
Brief Title: Percutaneous High Frequency Alternating Current Stimulation in Healthy Volunteers With 30kHz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neuromodest-pHFAC30
Record Dates: First submitted 2021-05-05; First posted 2021-05-13 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-05

CONDITIONS: Electrical Stimulation; Neuromodulation
Keywords: High-frequency alternating current; nerve block; somatosensory threshold; motor threshold; percutaneous electrical stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 kHz stimulation (Experimental): Percutaneous application of high frequency electrical current at 30 kHz over the median nerve for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
  Interventions: Device: 30 kHz stimulation (Myomed 932, Enraf-Nonius)
- Sham stimulation (Experimental): Electrodes are placed over the median nerve for 20 minutes in the same manner as experimental group but will be applied a sham electrical stimulation increasing the current intensity during the first 30 seconds.
  Interventions: Device: Sham stimulation (Myomed 932, Enraf-Nonius)

INTERVENTIONS:
Device: 30 kHz stimulation (Myomed 932, Enraf-Nonius) — A charge-balanced, symmetric, biphasic sinusoidal current without modulation will be delivered at a frequency of 30 kHz. The stimulation intensity will be defined as that sufficient to produce a "strong but comfortable" sensation, just below motor threshold, over the median nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft,Netherlands)
  Arms: 30 kHz stimulation
Device: Sham stimulation (Myomed 932, Enraf-Nonius) — Sham stimulation will be delivered at a frequency of 30 kHz only during the first 30 seconds.
  Arms: Sham stimulation

SUMMARY:
High-frequency alternating currents of greater than 1 kHz applied on peripheral nerves has been used in animal studies to produce a motor nerve block. It has been evidenced that frequencies higher than 5 kHz are necessary to produce a complete peripheral nerve block in primates, whose nerve thickness is more similar to humans.

DETAILED DESCRIPTION:
The previous studies with transcutaneous and percutaneous HFAC, suggest high-frequency stimulation (10 and 20 kHz) have an inhibitory effect over muscle strength and somatosensory threshold.

However, the 30 kHz frequency has never been applied, and the hypothesis is that it can produce a greater blockage at the sensitive level and be a more comfortable application for the patient. The purpose of the present work is to determine if a greater blockage of the sensory component of the nerve occurs with this frequency and is to reduce the amount of current intensity needed using a percutaneous approach by apply two acupuncture needles near the nerve as electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Ability to perform all clinical tests and understand the study process, as well as obtaining informed consent.
* Tolerance to the application of electrotherapy.
* That they have not diagnosed any pathology.
* They do not present a contraindication to puncture and / or the application of electric currents.

Exclusion Criteria:

* Neuromuscular disease.
* Epilepsy.
* Trauma, surgery or pain affecting the upper limb
* Osteosynthesis material in the upper limb.
* Diabetes.
* Cancer.
* Cardiovascular disease.
* Pacemaker or other implanted electrical device.
* Take any drug (NSAIDs, corticosteroids, antidepressants, analgesics, antiepileptics, ...) during the study and in the previous 7 days.
* Presence of tattoos or other external agent introduced into the treatment or assessment area.
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Latency of Antidromic median sensory nerve action potential | Baseline at 0 minutes
  The recording electrodes were placed on the second finger and the stimulus will be applied on the median nerve (above the elbow joint). The stimulus will consist of a train of 10 pulses (100 μs width), applied at supramaximal stimulation, presented at 1 Hz (DS7A, Digitimer Ltd). Latency will be registered with a specific software (Signal software, CED) and will be expressed in millisecond.
Amplitude of Antidromic median sensory nerve action potential | Baseline at 0 minutes
  The recording electrodes were placed on the second finger and the stimulus will be applied on the median nerve (above the elbow joint). The stimulus will consist of a train of 10 pulses (100 μs width), applied at supramaximal stimulation, presented at 1 Hz (DS7A, Digitimer Ltd). Peak-to-peak amplitude (PPA) will be registered with a specific software (Signal software, CED) and will be expressed in millivolts.
Tactile Threshold | Baseline at 0 minutes
  The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Pressure Pain Threshold | Baseline at 0 minutes
  The PPT will be measured with an algometer and will be expressed in Newtons
Muscle strength | Baseline at 0 minutes
  Muscle strength will be measured with a dynamometer and will be expressed in Kgs.
Tactile Threshold | During treatment at 15 minutes
  The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Pressure Pain Threshold | During treatment at 15 minutes
  The PPT will be measured with an algometer and will be expressed in Newtons
Latency Antidromic median sensory nerve action potential | Immediately after treatment at 20 minutes
  The recording electrodes were placed on the second finger and the stimulus will be applied on the median nerve (above the elbow joint). The stimulus will consist of a train of 10 pulses (100 μs width), applied at supramaximal stimulation, presented at 1 Hz (DS7A, Digitimer Ltd). Latency (NPL) will be registered with a specific software (Signal software, CED) and will be expressed in millisecond.
Amplitude Antidromic median sensory nerve action potential | Immediately after treatment at 20 minutes
  The recording electrodes were placed on the second finger and the stimulus will be applied on the median nerve (above the elbow joint). The stimulus will consist of a train of 10 pulses (100 μs width), applied at supramaximal stimulation, presented at 1 Hz (DS7A, Digitimer Ltd). Peak-to-peak amplitude (PPA) will be registered with a specific software (Signal software, CED) and will be expressed in millivolts.
Tactile Threshold | Immediately after treatment at 20 minutes
  The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Pressure Pain Threshold | Immediately after treatment at 20 minutes
  The PPT will be measured with an algometer and will be expressed in Newtons
Muscle strength | Immediately after treatment at 20 minutes
  Muscle strength will be measured with a dynamometer and will be expressed in Kgs.
Latency Antidromic median sensory nerve action potential | Immediately after treatment at 30 minutes
  The recording electrodes were placed on the second finger and the stimulus will be applied on the median nerve (above the elbow joint). The stimulus will consist of a train of 10 pulses (100 μs width), applied at supramaximal stimulation, presented at 1 Hz (DS7A, Digitimer Ltd). Latency will be registered with a specific software (Signal software, CED) and will be expressed in millisecond.
Amplitude Antidromic median sensory nerve action potential | Immediately after treatment at 30 minutes
  The recording electrodes were placed on the second finger and the stimulus will be applied on the median nerve (above the elbow joint). The stimulus will consist of a train of 10 pulses (100 μs width), applied at supramaximal stimulation, presented at 1 Hz (DS7A, Digitimer Ltd). Peak-to-peak amplitude (PPA) will be registered with a specific software (Signal software, CED) and will be expressed in millivolts.
Tactile Threshold | Immediately after treatment at 30 minutes
  The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Pressure Pain Threshold | Immediately after treatment at 30 minutes
  The PPT will be measured with an algometer and will be expressed in Newtons
Muscle strength | Immediately after treatment at 30 minutes
  Muscle strength will be measured with a dynamometer and will be expressed in Kgs.

SECONDARY OUTCOMES:
Baseline nerve temperature | Baseline at 0 minutes, at 15 minutes, immediately after treatment at 20 minutes, and immediately after treatment at 30 minutes
  Nerve temperature will be measured using a termodoppler (Celsius degrees)
Numerical Discomfort Rate Score | After the intervention at 35 minutes
  the possible discomfort caused by the interventions will be assess by a numerical rate score. The NRS consists of a scale from 0 (no discomfort) to 10 (worst possible discomfort)
Numerical Pain Rate Score | After the intervention at 35 minutes
  The NRS consists of a scale from 0 (no pain) to 10 (worst possible pain)
Number of participants with intervention-related adverse effects | After the intervention at 35 minutes
  The possible adverse effects caused by the interventions will be assess by a closed questionnaire, where the presence of any adverse effect would be qualified as 1 point and the negative presence of adverse effect as 0 point.
Blinding success | After the intervention at 35 minutes
  Blinding of subjects and researchers will be assessed using the Bang questionary. It will be the question after the intervention, "What type of treatment do you think you have received?" Will be asked, with 5 items: (1) "I firmly believe that I have received an experimental treatment"; (2) "I slightly believe that I have received an experimental treatment"; (3) "I strongly believe that I have received a placebo"; (4) "I slightly think I have received a placebo"; (5) "Don't know, don't answer.", Index where -1 is blinded and 1 is unblinded.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Avendaño-Coy, PhD, Study Director — Castilla-La Mancha University
Locations (1):
- Castilla-La Mancha University, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarez DM, Serrano-Munoz D, Fernandez-Perez JJ, Gomez-Soriano J, Avendano-Coy J. Effect of percutaneous electrical stimulation with high-frequency alternating currents at 30 kHz on the sensory-motor system. Front Neurosci. 2023 Feb 9;17:1048986. doi: 10.3389/fnins.2023.1048986. eCollection 2023. PMID 36845426